CLINICAL TRIAL: NCT00858546
Title: The Influence of Low Frequency Repetitive Transcranial Stimulation (r-TMS) Treatment on Motor and Cognitive Measurements in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Oren Cohen, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-6874-OC-CTIL
Record Dates: First submitted 2009-03-08; First posted 2009-03-10 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active repetitive transcranial Stimulation (Experimental): Active repetitive transcranial Stimulation
  Interventions: Device: Repetitive transcranial stimulation

INTERVENTIONS:
Device: Repetitive transcranial stimulation — Repetitive transcranial stimulation

SUMMARY:
The aim of the study is to test the effects of low frequency deep rTMS using the novel H-coil on the motor, affective and cognitive deficits in patients with Parkinson's disease (PD) and to establish its safety in this population.

The investigators anticipate to recruit 10 patients to an open pilot study. All patients will receive an active rTMS stimulation and will be given 12 treatment sessions, over a period of up to 4 weeks. Each of the 12 daily treatment sessions (lasting about 30 minutes each), will be consisted of 25 stimulation trains over the prefrontal cortex (20Hz trains, 2 seconds each with an inter-train interval of 20 seconds) and one train of 15 minutes at 1 Hz over the the motor cortex.

The following outcome measures will be taken prior to the treatment (screening visit), and at day 1, 10, 30, 60, and 90:

1. Unified Parkinson's Disease Rating Scale (UPDRS )
2. Clinical Global Impression of Severity (CGIS)
3. Pegboard test.
4. Tapping test
5. Up & Go test
6. Abnormal Involuntary Movement Scale (AIMS) Mood and affect Beck Depression Inventory (BDI) Cognition

1. Mini mental State examination (MMSE) 2. Digit forward and backward tests. 3. Word fluency. 4. Frontal Assessment Battery (FAB)

Side effects will be closely monitored by the researchers and will be promptly reported to the IRB

ELIGIBILITY:
Inclusion Criteria:

* PD patients aged 40 years or older, diagnosed as idiopathic PD according to the UK Brain Bank criteria, with Hoehn & Yahr stages II - IV while "off".
* Participants on antidepressants should be at least 2 months on stable therapy

Exclusion Criteria:

* Patients who have concomitant epilepsy, a history of seizure or heat convulsion or history of epilepsy in first degree relative.
* Patients on neuroleptics.
* Patients with dementia or any unstable medical disorder.
* History or current Unstable hypertension.
* History of head injury or neurosurgical interventions.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
* History of migraine or frequent or severe headaches.
* History of hearing loss.
* The presence of cochlear implants
* History of drug abuse or alcoholism.
* Pregnancy or not using a reliable method of birth control.
* Participation in current clinical study or clinical study within 30 days prior to this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS ) | 1 year

SECONDARY OUTCOMES:
CGIS, Pegboard test,Tapping test,Up & Go test, AIMS,BDI MMSE, Digit forward and backward, Word fluency, FAB | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel